CLINICAL TRIAL: NCT05161221
Title: Adductor Canal Block With Liposomal Bupivacaine (Exparel) Versus Femoral Nerve Catheter for Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Trial
Brief Title: Post Operative Pain Management Through Adductor Canal Block With Bupivacaine for ACL Reconstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sham21D.369
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pain, Postoperative; ACL
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Tablets; Naproxen; Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pre-operative femoral nerve catheter (Active Comparator): participants undergoing ACL reconstruction surgery will receive a femoral prior to their surgery
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Naproxen 500 Mg; Drug: Tylenol Pill; Procedure: Femoral Nerve Catheter
- Pre-operative adductor canal block with liposomal bupivacaine (Active Comparator): participants undergoing ACL reconstruction surgery will receive a nerve block using liposomal Bupivacaine (Exparel)
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Naproxen 500 Mg; Drug: Tylenol Pill; Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: OxyCODONE 5 mg Oral Tablet — Participants will receive 20 OxyCODONE 5 mg Oral Tablet post surgery for pain control
Drug: Naproxen 500 Mg — Participant will receive Naproxen 500 Mg post surgery for pain control
Drug: Tylenol Pill — Participants will be instructed to take up to 1000mg of Tylenol by mouth for pain control
Drug: Liposomal bupivacaine — Participants will receive pre-operative adductor canal block with liposomal bupivacaine (Exparel)
  Other Names: Exparel
  Arms: Pre-operative adductor canal block with liposomal bupivacaine
Procedure: Femoral Nerve Catheter — Participants will receive pre-operative femoral nerve catheter
  Other Names: Femoral Nerve Block
  Arms: Pre-operative femoral nerve catheter

SUMMARY:
Liposomal bupivacaine injectable suspension (Exparel), manufactured by Pacira Pharmaceuticals, is an FDA-approved, long-lasting nonopioid analgesic that is indicated for single-dose infiltration in adults to produce postsurgical local analgesia. Exparel's extended bioavailability allows for 48 hours of pain control. Periarticular infiltration of liposomal bupivacaine has been safely and effectively used for total knee arthroplasty as an alternative to FNBs, avoiding transient quadriceps weakness and potential in-hospital falls. Recently Exparel has been FDA approved for interscalene brachial plexus nerve block to produce postsurgical regional analgesia for upper extremity/shoulder procedures. It is not yet approved for peripheral nerve blocks of the lower extremity.

No study to date, to our knowledge, has evaluated the efficacy of single-dose adductor canal blockade with Exparel compared to femoral nerve catheter with bupivacaine. We pose that Exparel used for an adductor canal block can offer the benefit of a single-dose injection with extended pain control without the burden of an indwelling catheter and to avoid adverse events of femoral nerve blockade related to quadriceps weakness and dysesthesias.

The purpose of this study is to determine whether adductor canal blockade with liposomal bupivacaine (Exparel) is a safe and effective alternative to femoral nerve catheters for post-operative pain control for patients undergoing ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing primary anterior cruciate ligament reconstruction with autograft
2. Has not used narcotic pain medication in 3 months
3. Ages of 18+
4. Proficient in the English language
5. Willing and able to follow study protocol

Exclusion Criteria:

1. ACL repair, revision surgery, or allograft
2. Multi-ligamentous knee injuries
3. Cartilage procedures that prevented adherence to the immediate weightbearing and range of motion rehabilitation protocol
4. Patients taking baseline opioid for other injury
5. Dementia or other psychiatric illness that would preclude accurate evaluation
6. Pregnant or lactating patients
7. Non-English speakers as questionnaires are only available in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-12-06 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 8 weeks
  Participant will record Patient Satisfaction through Visual Analog Scale for pain
Post operative pain management | 8 weeks
  Participant will receive 20 5mg tablets of Oxycodone and will record opioid consumption through post operative instruction sheets from pain control regiments.
Post operative pain management | 8 weeks
  Participant will record quadriceps function tests

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States